CLINICAL TRIAL: NCT05587517
Title: A Clinical Trial of Interventions to Support Family Surrogates of Critically Ill Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-09023929; R01NR019831 (NIH)
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Grief; Trauma; Psychotherapy; Critical Care
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Mixed methods randomized controlled trial (RCT) to further evaluate the efficacy of EMPOWER for reducing surrogate symptoms of PTSD and PGD.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMPOWER arm (Experimental): The EMPOWER arm includes six 15 minute modules delivered in a 1-on-1 format with the same interventionist, and 2 boosters (approximately 45 minutes each) conducted by phone.
  Subjects who meet eligibility criteria will receive up to 4 sequential assessments before and after the EMPOWER intervention within 3 months conducted in person and by phone.
  Interventions: Behavioral: EMPOWER
- Supportive Conversation arm (Placebo Comparator): The Supportive Conversation (SC) arm includes a supportive, empathic encounter without specific skill-building for approximately the same amount of time as EMPOWER.
  Subjects who meet eligibility criteria will receive up to 4 sequential assessments before and after SC within 3 months conducted in person and by phone.
  Interventions: Other: Supportive Conversation

INTERVENTIONS:
Behavioral: EMPOWER — EMPOWER is a manualized treatment delivered based in cognitive behavioral and acceptance and commitment therapies delivered by a trained mental health professional that utilizes breathing and grounding exercises, mindfulness meditation, psychoeducation, imaginal dialogue with the patient, and coping rehearsal techniques.
  The total amount of time EMPOWER intervention is about 90 minutes, about 15 minutes each module. It can either be administered in one session or many sessions to accommodate the dynamic nature of ICU, and has two booster follow-up calls (roughly 45 minutes each) in the month following initial treatment.
  Arms: EMPOWER arm
Other: Supportive Conversation — The Supportive Conversation will match the time and attention offered through EMPOWER, so will be about 1.5-2 hours and will have two additional follow-up calls.
  Arms: Supportive Conversation arm

SUMMARY:
Hypotheses 1a and 1b: Compared to Supportive Conversation arm, the EMPOWER intervention will significantly decrease surrogate decision makers' symptoms of grief and Post Traumatic Stress Disorder (PTSD) (primary outcomes); and H1b. experiential avoidance, depression, regrets, and increases in patients' value-concordant care (secondary outcomes) at T1-T4.

Hypothesis 2. Qualitative data will provide insights not captured by quantitative data.

Hypothesis 3. Reductions in experiential avoidance will mediate reductions in grief and Post Traumatic Stress Disorder (PTSD) symptoms, highlighting it as important to target in future implementation.

DETAILED DESCRIPTION:
Intensive Care Units (ICUs) are stressful places fraught with grief for family members who witness dying loved ones, often in pain, struggling to breathe and/or maintain consciousness. Compounding their distress, family members are often thrust into the position of patient "surrogate," needing to make life-and-death decisions on the patient's behalf. Researchers have shown that end-of-life (EoL) decision-making is undermined by grief, which interferes with acceptance of the patient's impending death and leads to care choices that adversely affect patients' quality of care and death.1-3 These circumstances heighten surrogates' risk of meeting criteria for Prolonged Grief Disorder (PGD), Posttraumatic Stress Disorder (PTSD), and decisional regret about the EoL care that the patient received, each associated with poor bereavement outcomes.4-7 Nearly 60% of ICU surrogates report moderate to extreme grief; 34% report extreme levels of peritraumatic stress symptoms.1

The coronavirus (COVID-19) pandemic has made an already bad situation worse. At the start of the pandemic, social distancing policies forced millions of families to confront obstacles to communication, medical decision-making, and care.8-10 Surrogates were left struggling with severe pre-loss grief and peritraumatic stress -- intensely longing to be near to the patient, confused about their roles, lonely, horrified, angry, disoriented and emotionally numb.10,11 Now, as the Delta variant creates a new "wave" of mortality and infection, bereaved family members may have remorse about vaccine refusal,12 feel guilty for transmitting the virus to the patient, or regret decisions about EoL care. With over 35 million cases and 600,000 deaths in the United States from COVID-19,13 the need for psychosocial interventions to support surrogates in the ICU is clear.

Prior efforts to address the plight of family surrogates of critically ill patients have proved disappointing14-20 - with one ICU intervention significantly increasing the surrogate's severity of PTSD symptoms.14 A key limitation of these interventions is that while they targeted psychological outcomes, they were not psychological interventions. To address this, the investigators developed a brief, flexibly administered cognitive-behavioral, acceptance-based psychological intervention called EMPOWER (Enhancing & Mobilizing the POtential for Wellness & Emotional Resilience).21,22 Our pilot NIH-R21 (N=39) showed that EMPOWER had superior efficacy to enhanced usual care for reducing symptoms of PGD (d=1.20) and PTSD (d=.99). Consistent with mediation, EMPOWER reduced experiential avoidance (d=1.20); these reductions were correlated with PGD and PTSD change scores (p<0.01). Large reductions in decisional regret (d=1.57) were observed, with no notable differences by surrogate race or delivery format (telehealth vs. in-person).

Investigators propose to conduct a Phase II mixed methods randomized controlled trial (RCT) to further evaluate the efficacy of EMPOWER for reducing surrogate symptoms of PTSD and PGD. Surrogates (N=172) will be randomized to EMPOWER (n=86) or a standardized supportive conversation (SC; n=86). Effects of the intervention will be assessed via measures administered pre-intervention (T1), immediately post-intervention (T2), and at 3 months (T3), and 12 months (T4) following the T2 assessment. Investigators will also conduct semi-structured interviews with surrogates (n≈48) to probe intervention effects on mental health and explore contextual factors (e.g., medical mistrust, visitation restrictions) likely to affect surrogates during the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Patients who, during their hospital stay, have been admitted to the ICU and are near EoL, as indicated by a modified "surprise question" whereby physicians are asked to identify patients whom they do not expect to survive the next 12 months.
* Surrogate decision-makers of patients who were admitted to the ICU or step-down unit during their current admission/stay, or within 1 month of discharge from their last admission/stay.
* Surrogate decision-makers are 18 years or older.
* Surrogate decision-makers whom physicians or advance practice providers (i.e. physician assistants, nurse practitioners) indicate as the designated health care proxy or decision-making patient surrogates, or who are listed as such in the patient's medical charts or by self-report of the surrogate.
* Surrogate decision-makers must speak English.
* Surrogate decision-makers must report "syndromal" levels of pre-loss grief (PG-12 score ≥ 25) or peritraumatic distress (PDI ≥ 23).
* Surrogate decision makers will need to reside in a state in which an interventionist is licensed or otherwise be able to comply with current telehealth regulations.
* Surrogate decision-makers will need to be willing to utilize a device (computer, tablet, phone) with internet.
* Surrogate decision-makers who are able and willing to provide an emergency contact.

Exclusion Criteria:

* Patients and surrogate decision-makers who do not meet the eligibility criteria.
* Surrogate decision-makers who indicate the presence of cognitive impairment based on responses to the Ultra-Brief Confusion Assessment Method and/or significant psychiatric or cognitive disturbance sufficient, in the investigator/study staff's judgment, to preclude completion of the assessment measures, interview or informed consent.
* Surrogate-decision makers who endorse suicidal ideation in the past month based on responses to the Columbia Suicide Severity Rating Scale.
* Surrogate-decision makers who are unable to access a functional device for videoconferencing and decline the offer to use a study loner device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2027-12-11 (Estimated); Study Completion 2027-12-11 (Estimated)

PRIMARY OUTCOMES:
Change of Prolonged Grief Disorder | from baseline through twelve-month follow-up
  Symptoms of prolonged grief disorder, as measured by the Prolonged Grief-13-Revised, will be compared between the week following the intervention, at one month follow-up and at twelve-month follow-up . The PG-13-R consists of 13 items and total score can range from 0 to 62. Higher total scores represent greater symptom burden. Lower scores represent better outcomes.
Change of Post-Traumatic Stress Disorder | From baseline through twelve-month follow-up
  Symptoms of post-traumatic stress disorder, as measured by the Impact of Events Scale-Revised, will be compared between groups at baseline through twelve-month follow up assessments . The IES-R consists of 22 items and total score can range from 0 to 88. Higher total scores represent greater symptom burden. Lower scores represent better outcomes.
Change of Anticipatory Grief | from baseline through twelve-month follow-up
  Symptoms of anticipatory grief, as measured by the PG-12-R, consists of 12 items using a 5-point Likert scale. Total scores range from 11 to 55, with higher scores representing greater anticipatory grief.

SECONDARY OUTCOMES:
Change of Depression | From baseline through twelve-month follow-up
  Symptoms of depression, as measured by the Hospital Anxiety and Depression Scale (HADS), will be compared between groups at from baseline through twelve-month follow-up . HADS consists of 7 questions in their 14-item scale that assess depression. Higher scores indicate higher symptom burden. Lower scores represent a normal range.
Change of Regret | From baseline through twelve-month follow-up
  Regret, as measured by the Decision Regret Scale, will be compared between groups at baseline through twelve-month follow-up . The decision regret scale is a one-item likert-style measure. Total scores can range from 5 to 25. Higher total scores represent greater symptom burden. Lower scores represent better outcomes.
Change of Peritraumatic Distress | 1 week following the intervention through twelve-month follow-up .
  Symptoms of peritraumatic distress, as measured by the Peritraumatic Distress Inventory (adapted to fi the ICU experience), will be compared between groups in the week following the intervention through the twelve-month-follow up . The PDI consists of 13 likert-style items and total score can range from 0 to 52. Higher total scores represent greater symptom burden. Lower scores represent better outcomes.
Change of Anxiety | From baseline through twelve-month follow-up
  Symptoms of anxiety, as measured by the Hospital Anxiety and Depression Scale (HADS), will be compared between groups at from baseline through twelve-month follow-up ). HADS consists of 7 questions in their 14-item scale that assess anxiety. Higher scores indicate higher symptom burden. Lower scores represent a normal range.

OTHER OUTCOMES:
Change of Dissociation | From baseline to the 1 week following the intervention
  Symptoms of dissociation, as measured by the Peritraumatic Dissociative Experiences Questionnaire, will be compared between groups at baseline and the week following the intervention . The PDEQ consists of 10 items scored on a 5-point Likert scale. Scores range from 10 to 50, with higher scores representing greater symptoms of dissociation.
Change of Distress Tolerance | From baseline through twelve-month follow-up
  Symptoms of distress tolerance, as measured by the Distress Tolerance Short Form Scale, will be compared between groups at baseline through the twelve-month follow-up . The DTS-SF consists of four 5-point Likert items measuring the individual's perceived ability to experience and endure negative psychological states.
Change of Surrogate's Quality of Life | From the 1 week following the intervention through twelve-month follow-up
  Quality of life, as measured by Quality of Life/Death, will be compared between groups at the week following the intervention through the twelve-month follow-up . Scores range from 3 to 30, with lower scores representing better quality of life.
Satisfaction with Critical Care | At the three-month follow-up
  Satisfaction with critical care, as measured by Critical Care Family Satisfaction Survey, will be assessed at the three-month follow-up. The CCFSS-EMPOWER version consists of 12 items total, scored using a 1-5 Likert scale. Scores range from 12 to 60. Higher scores represent less satisfaction with care.
Patient's Symptoms | At baseline
  Surrogate-perceived Patient Symptoms consists of two items on 10-point Likert scale that measure surrogate-perceived patient symptoms of patient pain and dyspnea. This assessment will be administered at baseline by the. Scores range from 1 to 10 each, with higher scores representing greater surrogate-perceived pain or dyspnea.
Change of Patient's Quality of Death | From one-month to twelve-month follow-up
  Quality of Death will be measured using the Caregiver Evaluation of the Quality of End-of-Life Care (CEQUEL). Total score can range from 13 to 26. Higher total scores represent better caregiver-assessed patient quality of death. Higher total scores represent better outcomes.
Change of General Physical and General Mental Health | From baseline through twelve-month follow-up
  PROMIS-GH consists of 10-items, with each utilizing a 7-day recall period. The initial 9-items make us of a 5-point scale, with 3 separate verbal anchors that ask patients to rate their health or abilities, indicate how often they are experiencing a phenomenon or how severe their symptomatic experience is. The final item asks patients to indicate their pain on a 0-10 numeric rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Prigerson, PhD, Principal Investigator — Weill Medical College of Cornell University; Wendy Lichtenthal, PhD, Principal Investigator — University of Miami
Locations (3):
- United States (3):
  - University of Miami, Miami, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NewYork-Presbyterian Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
All participant data, including self-report measures and qualitative interviews, will be shared to qualified investigators under a Data Use Agreement in de-identifiable form. Data will be made available upon approval of PIs and will be used solely for research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available once the study's specific aims will be published and will be destroyed once analyses are completed.
Access Criteria: Accessing data requires making a formal request at the appropriate time and the PIs and investigative team will review the request. If approved, the data analyst from our Cornell Center for Research on End-of-Life Care will make a de-identifiable dataset to address the analyses in the request.

REFERENCES:
- [Background] Derry HM, Lief L, Schenck EJ, Berlin DA, Prigerson HG. Peritraumatic Stress among Caregivers of Patients in the Intensive Care Unit. Ann Am Thorac Soc. 2020 May;17(5):650-654. doi: 10.1513/AnnalsATS.201908-647RL. No abstract available. PMID 32068429
- [Background] Givens JL, Prigerson HG, Kiely DK, Shaffer ML, Mitchell SL. Grief among family members of nursing home residents with advanced dementia. Am J Geriatr Psychiatry. 2011 Jun;19(6):543-50. doi: 10.1097/JGP.0b013e31820dcbe0. PMID 21606897
- [Background] Maciejewski PK, Prigerson HG. Emotional numbness modifies the effect of end-of-life discussions on end-of-life care. J Pain Symptom Manage. 2013 May;45(5):841-7. doi: 10.1016/j.jpainsymman.2012.04.003. Epub 2012 Aug 25. PMID 22926093
- [Background] Siegel MD, Hayes E, Vanderwerker LC, Loseth DB, Prigerson HG. Psychiatric illness in the next of kin of patients who die in the intensive care unit. Crit Care Med. 2008 Jun;36(6):1722-8. doi: 10.1097/CCM.0b013e318174da72. PMID 18520637
- [Background] Wright AA, Keating NL, Balboni TA, Matulonis UA, Block SD, Prigerson HG. Place of death: correlations with quality of life of patients with cancer and predictors of bereaved caregivers' mental health. J Clin Oncol. 2010 Oct 10;28(29):4457-64. doi: 10.1200/JCO.2009.26.3863. Epub 2010 Sep 13. PMID 20837950
- [Background] Wright AA, Zhang B, Ray A, Mack JW, Trice E, Balboni T, Mitchell SL, Jackson VA, Block SD, Maciejewski PK, Prigerson HG. Associations between end-of-life discussions, patient mental health, medical care near death, and caregiver bereavement adjustment. JAMA. 2008 Oct 8;300(14):1665-73. doi: 10.1001/jama.300.14.1665. PMID 18840840
- [Background] Zhang B, Nilsson ME, Prigerson HG. Factors important to patients' quality of life at the end of life. Arch Intern Med. 2012 Aug 13;172(15):1133-42. doi: 10.1001/archinternmed.2012.2364. PMID 22777380
- [Background] Bronsther R. Visitor Restrictions During COVID-19 Pandemic May Impact Surrogate Medical Decision-Making. J Patient Exp. 2020 Aug;7(4):428-429. doi: 10.1177/2374373520938489. Epub 2020 Jun 30. No abstract available. PMID 33062852
- [Background] Greenberg JA, Basapur S, Quinn TV, Bulger JL, Glover CM, Shah RC. Psychological Symptoms Among Surrogates of Critically Ill Patients During and Before the COVID-19 Pandemic. Chest. 2021 Jun;159(6):2318-2320. doi: 10.1016/j.chest.2020.12.056. Epub 2021 Jan 12. No abstract available. PMID 33444615
- [Background] Lamas D. I'm on the Front Lines. I Have No Plan for This. The New York Times. March 24, 2020.
- [Background] Wood J. These Harvard scientists think we'll have to socially distance until 2022. World Economic Forum2020, April 20.
- [Background] Luisa Paul M. People who have lost their loved ones to covid-19 are getting vaccinated, Alabama doctor says. The Washington Post2021.
- [Background] Centers for Disease Control and Prevention. COVIDView: A Weekly Surveillance Summary of U.S. COVID-19 Activity. 2021; https://www.cdc.gov/coronavirus/2019-ncov/covid-data/covidview/index.html.
- [Background] Carson SS, Cox CE, Wallenstein S, Hanson LC, Danis M, Tulsky JA, Chai E, Nelson JE. Effect of Palliative Care-Led Meetings for Families of Patients With Chronic Critical Illness: A Randomized Clinical Trial. JAMA. 2016 Jul 5;316(1):51-62. doi: 10.1001/jama.2016.8474. Erratum In: JAMA. 2017 May 23;317(20):2134. doi: 10.1001/jama.2017.4298. PMID 27380343
- [Background] Cox C, Monk A. Minority caregivers of dementia victims: A comparison of Black and Hispanic families. Journal of Applied Gerontology. 1990;9(3):340-354.
- [Background] Curtis JR, Back AL, Ford DW, Downey L, Shannon SE, Doorenbos AZ, Kross EK, Reinke LF, Feemster LC, Edlund B, Arnold RW, O'Connor K, Engelberg RA. Effect of communication skills training for residents and nurse practitioners on quality of communication with patients with serious illness: a randomized trial. JAMA. 2013 Dec 4;310(21):2271-81. doi: 10.1001/jama.2013.282081. PMID 24302090
- [Background] Dionne-Odom JN, Ejem DB, Wells R, Azuero A, Stockdill ML, Keebler K, Sockwell E, Tims S, Engler S, Kvale E, Durant RW, Tucker RO, Burgio KL, Tallaj J, Pamboukian SV, Swetz KM, Bakitas MA. Effects of a Telehealth Early Palliative Care Intervention for Family Caregivers of Persons With Advanced Heart Failure: The ENABLE CHF-PC Randomized Clinical Trial. JAMA Netw Open. 2020 Apr 1;3(4):e202583. doi: 10.1001/jamanetworkopen.2020.2583. PMID 32282044
- [Background] Lautrette A, Darmon M, Megarbane B, Joly LM, Chevret S, Adrie C, Barnoud D, Bleichner G, Bruel C, Choukroun G, Curtis JR, Fieux F, Galliot R, Garrouste-Orgeas M, Georges H, Goldgran-Toledano D, Jourdain M, Loubert G, Reignier J, Saidi F, Souweine B, Vincent F, Barnes NK, Pochard F, Schlemmer B, Azoulay E. A communication strategy and brochure for relatives of patients dying in the ICU. N Engl J Med. 2007 Feb 1;356(5):469-78. doi: 10.1056/NEJMoa063446. PMID 17267907
- [Background] White DB, Angus DC, Shields AM, Buddadhumaruk P, Pidro C, Paner C, Chaitin E, Chang CH, Pike F, Weissfeld L, Kahn JM, Darby JM, Kowinsky A, Martin S, Arnold RM; PARTNER Investigators. A Randomized Trial of a Family-Support Intervention in Intensive Care Units. N Engl J Med. 2018 Jun 21;378(25):2365-2375. doi: 10.1056/NEJMoa1802637. Epub 2018 May 23. PMID 29791247
- [Background] White DB, Cua SM, Walk R, Pollice L, Weissfeld L, Hong S, Landefeld CS, Arnold RM. Nurse-led intervention to improve surrogate decision making for patients with advanced critical illness. Am J Crit Care. 2012 Nov;21(6):396-409. doi: 10.4037/ajcc2012223. PMID 23117903
- [Background] Lichtenthal WG, Viola M, Rogers M, Roberts KE, Lief L, Cox CE, Brewin CR, Xu JC, Maciejewski PK, Pan CX, Coats T, Ouyang DJ, Rabin S, Vaughan SC, Breitbart W, Marenberg ME, Prigerson HG. Development and preliminary evaluation of EMPOWER for surrogate decision-makers of critically ill patients. Palliat Support Care. 2022 Apr;20(2):167-177. doi: 10.1017/S1478951521000626. PMID 34233779
- [Background] Prigerson HG, Viola M, Brewin CR, Cox C, Ouyang D, Rogers M, Pan CX, Rabin S, Xu J, Vaughan S, Gordon-Elliot JS, Berlin D, Lief L, Lichtenthal WG. Enhancing & Mobilizing the POtential for Wellness & Emotional Resilience (EMPOWER) among Surrogate Decision-Makers of ICU Patients: study protocol for a randomized controlled trial. Trials. 2019 Jul 9;20(1):408. doi: 10.1186/s13063-019-3515-0. PMID 31288829
- [Background] Creswell JW, Plano Clark VL. Designing and conducting mixed methods research. 2nd ed. Los Angeles: SAGE Publications; 2011
- [Background] Creswell JW, Clark VLP. Designing and conducting mixed methods research. Sage publications; 2017.
- [Background] Palinkas LA. Qualitative and mixed methods in mental health services and implementation research. J Clin Child Adolesc Psychol. 2014;43(6):851-61. doi: 10.1080/15374416.2014.910791. PMID 25350675
- [Background] Palinkas LA, Horwitz SM, Green CA, Wisdom JP, Duan N, Hoagwood K. Purposeful Sampling for Qualitative Data Collection and Analysis in Mixed Method Implementation Research. Adm Policy Ment Health. 2015 Sep;42(5):533-44. doi: 10.1007/s10488-013-0528-y. PMID 24193818
- [Background] Fusch PI, Ness LR. Are we there yet? Data saturation in qualitative research. The qualitative report. 2015;20(9):1408.
- [Background] Tariq S, Woodman J. Using mixed methods in health research. JRSM Short Rep. 2013 May 7;4(6):2042533313479197. doi: 10.1177/2042533313479197. Print 2013 Jun. PMID 23885291
- [Background] Haydar SA, Strout TD, Bond AG, Han PK. Prognostic value of a modified surprise question designed for use in the emergency department setting. Clin Exp Emerg Med. 2019 Mar;6(1):70-76. doi: 10.15441/ceem.17.293. Epub 2019 Mar 28. PMID 30944292
- [Background] Chiambretto P, Moroni L, Guarnerio C, Bertolotti G. [Italian validation of the Prolonged Grief Disorder Questionnaire (PG-12)]. G Ital Med Lav Ergon. 2008 Jan-Mar;30(1 Suppl A):A105-10. Italian. PMID 18700485
- [Background] Jacobsen JC, Zhang B, Block SD, Maciejewski PK, Prigerson HG. Distinguishing symptoms of grief and depression in a cohort of advanced cancer patients. Death Stud. 2010 Mar;34(3):257-73. doi: 10.1080/07481180903559303. PMID 20953316
- [Background] Kiely DK, Prigerson H, Mitchell SL. Health care proxy grief symptoms before the death of nursing home residents with advanced dementia. Am J Geriatr Psychiatry. 2008 Aug;16(8):664-73. doi: 10.1097/JGP.0b013e3181784143. PMID 18669945
- [Background] Prigerson HG, Boelen PA, Xu J, Smith KV, Maciejewski PK. Validation of the new DSM-5-TR criteria for prolonged grief disorder and the PG-13-Revised (PG-13-R) scale. World Psychiatry. 2021 Feb;20(1):96-106. doi: 10.1002/wps.20823. PMID 33432758
- [Background] Prigerson HG, Horowitz MJ, Jacobs SC, Parkes CM, Aslan M, Goodkin K, Raphael B, Marwit SJ, Wortman C, Neimeyer RA, Bonanno GA, Block SD, Kissane D, Boelen P, Maercker A, Litz BT, Johnson JG, First MB, Maciejewski PK. Prolonged grief disorder: Psychometric validation of criteria proposed for DSM-V and ICD-11. PLoS Med. 2009 Aug;6(8):e1000121. doi: 10.1371/journal.pmed.1000121. Epub 2009 Aug 4. PMID 19652695
- [Background] Bunnell BE, Davidson TM, Ruggiero KJ. The Peritraumatic Distress Inventory: Factor structure and predictive validity in traumatically injured patients admitted through a Level I trauma center. J Anxiety Disord. 2018 Apr;55:8-13. doi: 10.1016/j.janxdis.2018.03.002. Epub 2018 Mar 9. PMID 29549879
- [Background] Guardia D, Brunet A, Duhamel A, Ducrocq F, Demarty AL, Vaiva G. Prediction of trauma-related disorders: a proposed cutoff score for the peritraumatic distress inventory. Prim Care Companion CNS Disord. 2013;15(1):PCC.12l01406. doi: 10.4088/PCC.12l01406. No abstract available. PMID 23724345
- [Background] Fick DM, Inouye SK, Guess J, Ngo LH, Jones RN, Saczynski JS, Marcantonio ER. Preliminary development of an ultrabrief two-item bedside test for delirium. J Hosp Med. 2015 Oct;10(10):645-50. doi: 10.1002/jhm.2418. Epub 2015 Sep 15. PMID 26369992
- [Background] Motyl CM, Ngo L, Zhou W, Jung Y, Leslie D, Boltz M, Husser E, Inouye SK, Fick D, Marcantonio ER. Comparative Accuracy and Efficiency of Four Delirium Screening Protocols. J Am Geriatr Soc. 2020 Nov;68(11):2572-2578. doi: 10.1111/jgs.16711. Epub 2020 Sep 15. PMID 32930409
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Smith A. Mobile Access 2010| Pew Internet & American Life Project. Pew Research Center's Internet & American Life Project. 2010.
- [Background] Smith A. Technology trends among people of color. Pew Internet & American Life Project. 2010.
- [Background] Campos-Castillo C, Anthony D. Racial and ethnic differences in self-reported telehealth use during the COVID-19 pandemic: a secondary analysis of a US survey of internet users from late March. J Am Med Inform Assoc. 2021 Jan 15;28(1):119-125. doi: 10.1093/jamia/ocaa221. PMID 32894772
- [Background] Torous J, Jan Myrick K, Rauseo-Ricupero N, Firth J. Digital Mental Health and COVID-19: Using Technology Today to Accelerate the Curve on Access and Quality Tomorrow. JMIR Ment Health. 2020 Mar 26;7(3):e18848. doi: 10.2196/18848. PMID 32213476
- [Background] Alcantara C, Li X, Wang Y, Canino G, Alegria M. Treatment moderators and effectiveness of Engagement and Counseling for Latinos intervention on worry reduction in a low-income primary care sample. J Consult Clin Psychol. 2016 Nov;84(11):1016-1022. doi: 10.1037/ccp0000146. Epub 2016 Sep 15. PMID 27631958
- [Background] Martinez M, Perle JG. Reaching the Latino Population: a Brief Conceptual Discussion on the Use of Telehealth to Address Healthcare Disparities for the Large and Growing Population. Journal of Technology in Behavioral Science. 2019;4(3):267-273.
- [Background] Bartholomew TT, Lockard AJ. Mixed methods in psychotherapy research: A review of method(ology) integration in psychotherapy science. J Clin Psychol. 2018 Oct;74(10):1687-1709. doi: 10.1002/jclp.22653. Epub 2018 Jun 13. PMID 29900532
- [Background] Morse JM. "Data were saturated . . . ". Qual Health Res. 2015 May;25(5):587-8. doi: 10.1177/1049732315576699. No abstract available. PMID 25829508
- [Background] Brunet A, Weiss DS, Metzler TJ, Best SR, Neylan TC, Rogers C, Fagan J, Marmar CR. The Peritraumatic Distress Inventory: a proposed measure of PTSD criterion A2. Am J Psychiatry. 2001 Sep;158(9):1480-5. doi: 10.1176/appi.ajp.158.9.1480. PMID 11532735
- [Background] Gamez W, Chmielewski M, Kotov R, Ruggero C, Suzuki N, Watson D. The brief experiential avoidance questionnaire: development and initial validation. Psychol Assess. 2014 Mar;26(1):35-45. doi: 10.1037/a0034473. Epub 2013 Sep 23. PMID 24059474
- [Background] Gamez W, Chmielewski M, Kotov R, Ruggero C, Watson D. Development of a measure of experiential avoidance: the Multidimensional Experiential Avoidance Questionnaire. Psychol Assess. 2011 Sep;23(3):692-713. doi: 10.1037/a0023242. PMID 21534697
- [Background] Gough K, Hudson P. Psychometric properties of the Hospital Anxiety and Depression Scale in family caregivers of palliative care patients. J Pain Symptom Manage. 2009 May;37(5):797-806. doi: 10.1016/j.jpainsymman.2008.04.012. Epub 2008 Sep 11. PMID 18789643
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Background] Higgins PC, Garrido MM, Prigerson HG. Factors Predicting Bereaved Caregiver Perception of Quality of Care in the Final Week of Life: Implications for Health Care Providers. J Palliat Med. 2015 Oct;18(10):849-57. doi: 10.1089/jpm.2015.29001.hp. Epub 2015 Jul 17. PMID 26186021
- [Background] Mack JW, Weeks JC, Wright AA, Block SD, Prigerson HG. End-of-life discussions, goal attainment, and distress at the end of life: predictors and outcomes of receipt of care consistent with preferences. J Clin Oncol. 2010 Mar 1;28(7):1203-8. doi: 10.1200/JCO.2009.25.4672. Epub 2010 Feb 1. PMID 20124172
- [Background] Marmar CR, Weiss DS, Metzler TJ. The peritraumatic dissociative experiences questionnaire. In: Wilson JP, Keane TM, eds. Assessing psychological trauma and PTSD. New York, NY: The Guilford Press; 1997:412-428.
- [Background] Weiss DS, Marmar CR. The Impact of Event Scale - Revised. In: Wilson J, Keane TM, eds. Assessing psychological trauma and PTSD. New York: Guildford; 1996:399-411.
- [Background] Garner LE, Van Kirk N, Tifft ED, Krompinger JW, Mathes BM, Fraire M, Falkenstein MJ, Brennan BP, Crosby JM, Elias JA. Validation of the distress tolerance scale-short form in obsessive compulsive disorder. J Clin Psychol. 2018 Jun;74(6):916-925. doi: 10.1002/jclp.22554. Epub 2017 Nov 15. PMID 29139125
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809
- [Background] George LS, Breitbart W, Prigerson HG. "My Family Wants Something Different": Discordance in Perceived Personal and Family Treatment Preference and Its Association With Do-Not-Resuscitate Order Placement. J Oncol Pract. 2019 Nov;15(11):e942-e947. doi: 10.1200/JOP.19.00250. Epub 2019 Sep 11. PMID 31509484
- [Background] Jabbarian LJ, Maciejewski RC, Maciejewski PK, Rietjens JAC, Korfage IJ, van der Heide A, van Delden JJM, Prigerson HG. The Stability of Treatment Preferences Among Patients With Advanced Cancer. J Pain Symptom Manage. 2019 Jun;57(6):1071-1079.e1. doi: 10.1016/j.jpainsymman.2019.01.016. Epub 2019 Feb 19. PMID 30794935
- [Background] Ratshikana-Moloko M, Ayeni O, Tsitsi JM, Wong ML, Jacobson JS, Neugut AI, Sobekwa M, Joffe M, Mmoledi K, Blanchard CL, Mapanga W, Ruff P, Cubasch H, O'Neil DS, Balboni TA, Prigerson HG. Spiritual Care, Pain Reduction, and Preferred Place of Death Among Advanced Cancer Patients in Soweto, South Africa. J Pain Symptom Manage. 2020 Jul;60(1):37-47. doi: 10.1016/j.jpainsymman.2020.01.019. Epub 2020 Feb 8. PMID 32045675
- [Background] Tergas AI, Prigerson HG, Shen MJ, Bates LM, Neugut AI, Wright JD, Maciejewski PK. Latino Ethnicity, Immigrant Status, and Preference for End-of-Life Cancer Care. J Palliat Med. 2019 Jul;22(7):833-837. doi: 10.1089/jpm.2018.0537. Epub 2019 Apr 11. PMID 30973302
- [Background] Johnson JG, Zhang B, Greer JA, Prigerson HG. Parental control, partner dependency, and complicated grief among widowed adults in the community. J Nerv Ment Dis. 2007 Jan;195(1):26-30. doi: 10.1097/01.nmd.0000252009.45915.b2. PMID 17220736
- [Background] Mack JW, Block SD, Nilsson M, Wright A, Trice E, Friedlander R, Paulk E, Prigerson HG. Measuring therapeutic alliance between oncologists and patients with advanced cancer: the Human Connection Scale. Cancer. 2009 Jul 15;115(14):3302-11. doi: 10.1002/cncr.24360. PMID 19484795
- [Background] Balboni TA, Prigerson HG, Balboni MJ, Enzinger AC, VanderWeele TJ, Maciejewski PK. A scale to assess religious beliefs in end-of-life medical care. Cancer. 2019 May 1;125(9):1527-1535. doi: 10.1002/cncr.31946. Epub 2019 Mar 2. PMID 30825390
- [Background] LaVeist TA, Nickerson KJ, Bowie JV. Attitudes about racism, medical mistrust, and satisfaction with care among African American and white cardiac patients. Med Care Res Rev. 2000;57 Suppl 1:146-61. doi: 10.1177/1077558700057001S07. PMID 11092161
- [Background] Tekeste M, Hull S, Dovidio JF, Safon CB, Blackstock O, Taggart T, Kershaw TS, Kaplan C, Caldwell A, Lane SB, Calabrese SK. Differences in Medical Mistrust Between Black and White Women: Implications for Patient-Provider Communication About PrEP. AIDS Behav. 2019 Jul;23(7):1737-1748. doi: 10.1007/s10461-018-2283-2. PMID 30264207
- [Background] Gentzler ER, Derry H, Ouyang DJ, Lief L, Berlin DA, Xu CJ, Maciejewski PK, Prigerson HG. Underdetection and Undertreatment of Dyspnea in Critically Ill Patients. Am J Respir Crit Care Med. 2019 Jun 1;199(11):1377-1384. doi: 10.1164/rccm.201805-0996OC. PMID 30485121
- [Background] Higgins PC, Prigerson HG. Caregiver evaluation of the quality of end-of-life care (CEQUEL) scale: the caregiver's perception of patient care near death. PLoS One. 2013 Jun 6;8(6):e66066. doi: 10.1371/journal.pone.0066066. Print 2013. PMID 23762467
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Wasser T, Matchett S. Final version of the Critical Care Family Satisfaction Survey questionnaire. Crit Care Med. 2001 Aug;29(8):1654-5. doi: 10.1097/00003246-200108000-00038. No abstract available. PMID 11505160
- [Background] Schafer JL, Olsen MK. Multiple Imputation for Multivariate Missing-Data Problems: A Data Analyst's Perspective. Multivariate Behav Res. 1998 Oct 1;33(4):545-71. doi: 10.1207/s15327906mbr3304_5. PMID 26753828
- [Background] Raudenbush SW, Chan WS. Application of a hierarchical linear model to the study of adolescent deviance in an overlapping cohort design. J Consult Clin Psychol. 1993 Dec;61(6):941-51. doi: 10.1037//0022-006x.61.6.941. PMID 8113495
- [Background] Singer JD, Willett JB. Modeling the days of our lives: Using survival analysis when designing and analyzing longitudinal studies of duration and the timing of events. Psychol Bul. 1991;110:268-290.
- [Background] Clarke V, Braun V. Thematic analysis. J Posit Psychol. 2017;12(3):297-298.
- [Background] Cheong J. Accuracy of Estimates and Statistical Power for Testing Meditation in Latent Growth Curve Modeling. Struct Equ Modeling. 2011;18(2):195-211. doi: 10.1080/10705511.2011.557334. Epub 2011 Nov 14. PMID 27547021
- [Background] Muthén B, Asparouhov T. Causal effects in mediation modeling: An introduction with applications to latent variables. J Structural Equation Modeling: A Multidisciplinary Journal. 2015;22(1):12-23.
- [Background] Kraemer HC. Messages for Clinicians: Moderators and Mediators of Treatment Outcome in Randomized Clinical Trials. Am J Psychiatry. 2016 Jul 1;173(7):672-9. doi: 10.1176/appi.ajp.2016.15101333. Epub 2016 Mar 17. PMID 26988629
- [Background] Falzarano F, Prigerson HG, Maciejewski PK. The Role of Advance Care Planning in Cancer Patient and Caregiver Grief Resolution: Helpful or Harmful? Cancers (Basel). 2021 Apr 20;13(8):1977. doi: 10.3390/cancers13081977. PMID 33924214